CLINICAL TRIAL: NCT01814423
Title: Pharmacokinetic Study of Multi-dose Chloroquine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bandim Health Project (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-CQ
Record Dates: First submitted 2013-03-16; First posted 2013-03-20 (Estimated); Last update posted 2014-03-11 (Estimated); Status verified 2014-03

CONDITIONS: Malaria
Keywords: Plasmodium falciparum; malaria; chloroquine; pharmacokinetic; children
MeSH Terms: conditions — Malaria; Malaria, Falciparum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chloroquine-base 50 mg (Experimental): Chloroquine-base 10 mg/kg twice a day for 2 days and 5 mg/kg twice a day for another day.
  Interventions: Drug: Chloroquine-base 50 mg
- Chloroquine-base 70 mg (Active Comparator): Chloroquine-base 10 mg/kg twice a day for 2 days and 5 mg/kg twice a day for another 3 days.
  Interventions: Drug: Chloroquine-base 70 mg

INTERVENTIONS:
Drug: Chloroquine-base 50 mg
  Arms: Chloroquine-base 50 mg
Drug: Chloroquine-base 70 mg
  Arms: Chloroquine-base 70 mg

SUMMARY:
Chloroquine (CQ) remains an alternative cheap, safe and widely available drug. Our previous research has shown that double (50 mg/kg) standard dose CQ given in split doses had a 95% efficacy and was well tolerated and safe. Still, safety could be an issue when the dose of CQ is increased. Severe adverse events are caused by high peak concentrations of CQ. Using split doses of CQ avoids high peak concentrations enabling the safe administration of high doses, however, pharmacokinetic data are lacking.

Children included in the study will be given 50 mg/kg as split doses over 3 days or 70 mg/kg as split doses over 5 days. Treatment will be observed. Drug concentrations and adverse events will be monitored. On day 1, children and their mother/guardian will be requested to stay at the health centre between 9 am and 6 pm.

Fifteen children aged 2-10 years with uncomplicated P. falciparum malaria and fulfilling the inclusion criteria will be recruited into each study arm.

Following the end of treatment, the children will be seen on the morning of day 7, 14, 21 and 28.

Any child wishing to withdraw during the treatment phase and any child with reparasitaemia during the follow up will be given rescue treatment with arthemeter-lumefantrine or quinine according to treatment guidelines in Guinea-Bissau.

Final analysis will include a description of included children, proportions of adverse events and any serious adverse events, drug concentrations and their relation to adverse events, the proportion of children withdrawn or lost to follow up, the cumulative PCR corrected and uncorrected success and failure rates on day 28 and the proportion of early, late clinical and late parasitological treatment failures.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 2 years and < 10 years.
* Mono-infection with P. falciparum detected by microscopy. Parasitemia of 1.000-100.000/µl asexual forms.
* Axillary temperature ≥ 37.5 ˚C or a history of fever within 24 hours.
* Ability to swallow oral medication.
* Ability and willingness to comply with the study protocol.
* Informed consent from a parent or guardian

Exclusion Criteria:

* Signs or symptoms of severe malaria.
* Presence of general danger signs in children under 5.
* Persistent vomiting.
* Presence of severe malnutrition.
* Any evidence of chronic disease or acute infection other than malaria.
* Regular medication which may interfere with antimalarial pharmacokinetics.
* History of hypersensitivity reactions or contraindications to chloroquine.

Ages: 2 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2013-04; Primary Completion 2014-02 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Chloroquine serum concentration | Twice daily during treatment, on day 1 an additional 8 measurements.
  Filterpaper blood samples will be collected in the morning and evening on the days of treatment. On day 1 hourly during daytime.

SECONDARY OUTCOMES:
Parasitemia | Twice a day dúring treatment and then weekly until day 28.
  Blood smear for microscopy will be performed in the morning and evening on the days of treatment, and for the 50 mg group on day 3. During follow-uo weekly until day 28.

OTHER OUTCOMES:
Haemoglobin level | On day 0, 3 and 28.
  The haemoglobin level will be measured on the the specified days.
Blood pressure | On day 1 and day 28
  Will be measures on day 1 at midday and on day 28.
ECG | Will be measures on day 1 and on last treatment day.

CONTACTS AND LOCATIONS:
Overall Officials: Poul-Erik Kofoed, Ph.d, Principal Investigator — Bandim Health Project
Locations (1):
- Projecto de Saúde de Bandim, Bissau, Guinea-Bissau

REFERENCES:
- [Derived] Ursing J, Rombo L, Eksborg S, Larson L, Bruvoll A, Tarning J, Rodrigues A, Kofoed PE. High-Dose Chloroquine for Uncomplicated Plasmodium falciparum Malaria Is Well Tolerated and Causes Similar QT Interval Prolongation as Standard-Dose Chloroquine in Children. Antimicrob Agents Chemother. 2020 Feb 21;64(3):e01846-19. doi: 10.1128/AAC.01846-19. Print 2020 Feb 21. PMID 31907183